CLINICAL TRIAL: NCT05632575
Title: The Virtual Promotoras (VIP) Program for Young Latina Women: Testing the Feasibility of an eHealth Intervention to Promote Sexual Health Among Young Latina Women in the US South
Brief Title: The Virtual Promotoras Study: eHealth Intervention to Promote Sexual Health Among Young Latina Women in the US South
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-08-2646
Record Dates: First submitted 2022-11-04; First posted 2022-11-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Latinas; U.S. South; sexual health; healthcare access; mHealth

STUDY DESIGN:
Intervention Model Description: Observational, single group, pre-post test design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm: Virtual Promotoras Intervention (Other): Single-arm study. Pre and post intervention. Observational. Behavioral
  Interventions: Behavioral: Virtual Promotoras Program

INTERVENTIONS:
Behavioral: Virtual Promotoras Program — Participants will receive a unique participant code from the virtual promotoras (i.e., patient educators and navigators), to access the VIP mobile phone app intervention. This will give them access to the three main components of the VIP intervention:
  1. Educational Modules (8 evidence-based educational modules made by the VPs),
  2. Sexual and Reproductive Health Plan (SRHP): Quiz-style instrument to help the participant set goals for her sexual health and develop a set of questions to ask her provider.
  3. Virtual Promotora's (VP) chat room.: Opportunity for participant to ask any questions that she may have about sexual health (SH) or sexual healthcare access (SHCA), refine her SRHP. The VP will also help her make her appointment for her clinical visit with one of the local free clinics which do not require insurance and are youth-friendly, and practice having the conversation that she wants to have with her clinical provider.

SUMMARY:
Young Latina women face significant barriers to sexual health and healthcare access, particularly in emerging Latino states like Alabama. The goals of the proposed study are to develop and examine the feasibility of an innovative, scalable mHealth, "safe space" intervention for Young Latina Women (YLW) in Alabama (AL) and to stimulate the conduct of behavioral research at the University of Alabama. This work is consistent with the National Institute of Nursing Research's goals of "Enhancing wellness by understanding the physical, behavioral, cultural and environmental influences on health status and developing culturally tailored interventions to prevent illness and promote health" and "Using innovative technologies to develop novel interventions that deliver personalized care and real-time health information to patients, families and healthcare providers".

DETAILED DESCRIPTION:
The goals of the proposed study are to develop and examine the feasibility of an innovative, scalable mHealth, "safe space" intervention for Young Latina Women (YLW) in Alabama (AL) and to stimulate the conduct of behavioral research at the University of Alabama (UA). YLW are disproportionately affected by sexual health (SH) disparities compared to their non-Hispanic White counterparts. In 2017, the birth rate for AL Latinas, 15-19 years of age, was 52.5/1,000 population compared to 22.9 among their non-Hispanic white counterparts. In 2016, the estimated rate of Hispanics living with diagnosed HIV infection in AL was 285.0/100,000 compared to 124.9/100,000 for non-Hispanic Whites. Forty-six percent of AL youth, in grades 9-12th, report having initiated sexual intercourse. Sexually active adolescents 15 years and older should be regularly screened for sexually transmitted infections (STI) and therefore must have access to healthcare services, timely screenings and (when desired) contraception to adequately care for their SH and make informed SH choices. However, Hispanic youth are significantly less likely than their non-Hispanic Black and non-Hispanic white counterparts to have a usual place for preventive care. Additionally, evidence-based, culturally relevant SH education programming is largely unavailable AL. There is a need for accessible, effective and scalable SH and sexual healthcare access (SHCA) interventions for YLW. The Virtual Promotoras Program (VIP) seeks to address this need.

The VIP is centered on the principle that creating a virtual "safe space" for YLW to learn about SH and SHCA can help them become more empowered to effectively care for their SH (i.e., develop reproductive health goals and plans), engage with the healthcare system (i.e., make and keep medical appointments, effectively communicate with provider etc.) and acquire needed preventive services. These strategies have been shown to improve health outcomes and reduce health disparities among adolescents, including Latino/a/x youth.

Extensive formative work conducted in 2017-2018 (44 semi-structured qualitative interviews with YLW, Latino/a/x parents, sexual healthcare providers and other key stakeholders) with active engagement of the Latino/a/x community and guided by a Community Based Participatory Research (CBPR) philosophical framework identified the following themes: lack of SH education in schools; lack of awareness of available sexual healthcare services and how to navigate them; embarrassment or lack of confidence in accessing sexual healthcare; and a desire to learn about SH and healthcare access through technology. This intervention development study is based on that research. Intervention mapping was used to create a detailed intervention outline for the VIP and design a promotoras' (peer navigator) capacity building training and manual.

This study includes the development and feasibility of the proposed mHealth VIP Program, which, if successful, will inform a large-scale randomized trial. Social Cognitive Theory, which postulates that cognitive, behavioral and environmental factors determine human behavior, guides this work. The mHealth VIP tool (mobile app) will create a virtual "safe space" where YLW can: learn about SH and SHCA (educational modules); connect with "virtual promotoras" who can provide guidance and advice on how to navigate the healthcare system (e.g. where to get services if you are uninsured); and create a SH plan (i.e., a goal setting and patient/provider communication tool). mHealth interventions show great promise toward increasing health-seeking behaviors, including SHCA among young populations. A majority of YLW have smartphones and half report being online "almost constantly", making mHealth interventions a natural choice for health promotion among this group. Reproductive/SH plans and patient-provider communication checklists are cost-effective but underutilized tools with potential to improve SH outcomes among YLW. Additionally, the literature on adult Latinas, shows that patient navigation is effective at linking Latinas to healthcare services. However, no other researchers in the US South are working with YLW to develop evidence-based SH education and peer navigator model to increase SH and SHCA empowerment and decrease SH disparities in this group. The specific aims of this study are: (1) Develop and examine the feasibility of a theory-based, culturally relevant SH and SHCA intervention for YLW; and (2) Estimate the parameters required to size a group randomized trial for the evaluation of efficacy of the VIP program. This work is consistent with the National Institute of Nursing Research's goals of "Enhancing wellness by understanding the physical, behavioral, cultural and environmental influences on health status and developing culturally tailored interventions to prevent illness and promote health" and "Using innovative technologies to develop novel interventions that deliver personalized care and real-time health information to patients, families and healthcare providers". This R15 will help grow the research enterprise at UA and provide unique and previously unavailable research opportunities to UA undergraduate, graduate and medical education students.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be eligible to participate if they self-identify as Latina, are 16-21 years of age, self-report not having had a preventive care or sexual healthcare visit in the last 18 months, and have lived in AL for at least 5 years.

Exclusion Criteria:

* Non-English or Spanish Speaking. (At this time, we are unable to accommodate Latinas who only speak indigenous languages.)

Ages: 16 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
sexual health and healthcare access empowerment | 3 months
  The main goal of the proposed intervention is to develop and evaluate the feasibility of a culturally relevant, evidence based sexual health education (knowledge and skill building) and healthcare intervention to empower YLW to care for their SH and make informed reproductive health choices9. This is a development and feasibility study; therefore an evaluation of effectiveness of the intervention will not take place at this point. However, the key outcomes of the intervention are SH empowerment and SHCA empowerment.
  The Sexual and Reproductive Empowerment (SRE) for Adolescents and Young Adults Scale, developed by Upadhyay and colleagues (2021) will be utilized to measure this outcome. The scale includes 95 items in 3 subscales: Access to sexual and reproductive information; Access to sexual and reproductive health services; and use of Desired contraceptive method. Items are measured on a 5-point Likert scale from "not at all true" to "extremely true".

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Alabama, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No